CLINICAL TRIAL: NCT05230537
Title: A Randomized, Participant and Investigator Masked, Placebo-controlled, Multicenter, Proof-of-concept Study to Assess the Safety and Efficacy of LNP023 (Iptacopan) in Patients With Early and Intermediate Age-related Macular Degeneration
Brief Title: A Masked, Placebo-controlled Study to Assess Iptacopan in Age-related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNP023E12201; 2021-001797-31 (EudraCT Number)
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; Macular degeneration; vision loss, macula damage; retina damage; dry macular degeneration; wet macular degeneration; AMD; Best Corrected Visual Acuity; Neovascular AMD; OCT
MeSH Terms: conditions — Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration | interventions — iptacopan

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, participant and investigator masked, placebo controlled, proof-of-concept study to assess the safety and efficacy of LNP023 in participants with early to intermediate age-related macular degeneration (e/iAMD) in one eye and neovascular age-related macular degeneration (nAMD) in the other eye.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigator and Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iptacopan (LNP023) (Experimental): Iptacopan (LNP023) oral use capsules
  Interventions: Drug: Iptacopan (LNP023)
- Placebo (Placebo Comparator): Placebo matched to study drug, oral use capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iptacopan (LNP023) — oral capsules
  Arms: Iptacopan (LNP023)
Drug: Placebo — oral capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of Iptacopan to prevent conversion of early or intermediate age-related macular degeneration (AMD) eyes to new incomplete retinal pigment epithelium and outer retinal atrophy (iRORA) or late AMD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, participant and investigator masked, placebo controlled, proof-of-concept study to assess the safety and efficacy of Iptacopan (LNP023) in participants with early to intermediate age-related macular degeneration in one eye and neovascular age-related macular degeneration in the other eye. All enrolled participants must have early/intermediate AMD in one eye, with at least one high risk optical coherence tomography (OCT) feature (study eye) and neovascular AMD in the other eye (fellow eye).

Participants who meet all of the eligibility criteria will be randomized at the Baseline/Day 1 visit in a 1:1 ratio into one of two treatment arms:

* Iptacopan (LNP023) oral capsules
* Placebo oral capsules Approximately 146 participants (73 per arm) will be treated worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥ 50 years of age
* Diagnosis of early or intermediate age-related macular degeneration (AMD) in the study eye as determined by the investigator on fundus examination
* Study eye (early/intermediate AMD eye) must have at least one high risk optical coherence tomography (OCT) feature (as defined by a central reading center).
* Diagnosis of neovascular AMD (nAMD) in the fellow eye as determined by the investigator.
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infection are required prior to the start of the treatment with LNP023.
* If not received previously, vaccination against Haemophilius influenzae infection should be given, if available and according to local regulations.

Exclusion Criteria:

* History or current diagnosis of ECG abnormalities indicating significant safety risk, such as clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia and clinically significant second or third degree atrioventricular block (AV block) without a pacemaker.
* History of familial long QT syndrome or known family history of Torsades de Pointes
* History of stroke or myocardial infarction during the 6-month period prior to Baseline/Day 1, any current clinically significant arrhythmias, or any advanced cardiac or severe pulmonary hypertension
* History of end stage kidney disease requiring dialysis or renal transplant
* History of malignancy of any organ system
* History of solid organ or bone marrow transplantation
* History of recurrent meningitis or history of meningococcal infections despite vaccination
* History of immunodeficiency diseases, including a positive Human Immunodeficiency Virus test result at Screening
* Active Hepatitis B (HBV) or Hepatitis C (HCV) infection
* History of hypersensitivity to any of the study treatments or excipients or to drugs of similar chemical classes or clinically relevant sensitivity to fluorescein dye as assessed by the Investigator.
* Evidence of cRORA or exMNV in the study eye based on multimodal imaging as determined by the central reading center.
* Participants who have current active TB as evidenced by clinical, radiographic and laboratory tests.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Development of new incomplete retinal pigment epithelium & outer retinal atrophy or late age-related macular degeneration (AMD) in the early/intermediate AMD eye as determined by optical coherence tomography (OCT) & supported by multimodal imaging | Baseline/Day 1 through Month 24
  OCT and other imaging will be performed using spectral domain OCT or swept source OCT machines

SECONDARY OUTCOMES:
The incidence of ocular and non-ocular adverse events (AEs) | Baseline/Day 1 through Month 24
  An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Change in Early Treatment Diabetic Retinopathy Study (ETDRS) (Standard Luminance) best corrected visual acuity (BCVA) scores in the early/intermediate AMD eye | Baseline/Day 1 through Month 24
  Best corrected visual acuity (BCVA) will be measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart. The number of letters read correctly, for each eye, will be recorded. Participants at sites in some countries may conduct BCVA testing using numerical charts rather than letter charts.
Change in ETDRS low luminance visual acuity (LLVA) scores in the early/intermediate AMD eye | Baseline/Day 1 through Month 24
  ETDRS low luminance visual acuity (LLVA) scores will be measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart. The number of letters read correctly, for each eye, will be recorded. Participants at sites in some countries may conduct BCVA testing using numerical charts rather than letter charts.
Change in contrast sensitivity (CS) scores in the early/intermediate AMD eye | Baseline/Day 1 through Month 24
  Pelli-Robson contrast sensitivity measurements will be performed using a Pelli-Robson contrast sensitivity wall chart and recording the number of correct letters read.
Change in Standard luminance manifold contrast vision meter contrast sensitivity (MCVM-CS) scores in the early/intermediate AMD eye | Baseline/Day 1 through Month 24
  MCVM contrast sensitivity measurements will be performed using an automated device that uses an adaptive algorithm to rapidly measure a contrast sensitivity function in 5-10 minutes.
Pharmacokinetics - concentrations of LNP023 related to trough samples | Baseline/Day 1 through Month 24
  Bioanalytical determination of plasma LNP023 concentrations related to trough samples using a LC-MS (mass spectrometry) method.
Change in low luminance manifold contrast vision meter (MCVM) contrast sensitivity scores in the early/intermediate AMD eye | Baseline/Day 1 through Month 24
  MCVM contrast sensitivity measurements will be performed using an automated device that uses an adaptive algorithm to rapidly measure a contrast sensitivity function in 5-10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (22):
  - Retina Consultants of Orange County, Fullerton, California
  - Salehi Retina Institute, Huntington Beach, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Southwest Retina Research Center, Durango, Colorado
  - Advanced Research LLC, Deerfield Beach, Florida
  - Retina Center Of South Florida, Delray Beach, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina Associates New Orleans, New Orleans, Louisiana
  - Retina Care Center, Baltimore, Maryland
  - Opthamalic Consultants of Boston, Boston, Massachusetts
  - Envision Ocular LLC, Bloomfield, New Jersey
  - Duke Eye Center, Durham, North Carolina
  - Retina Northwest PC, Portland, Oregon
  - Charles Retina Institute, Germantown, Tennessee
  - Austin Research Center for Retina, Austin, Texas
  - Retina Consultants TX Rsrch Ctr, Bellaire, Texas
  - Retina Foundation, Dallas, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Retina Consultants of Houston PA, Houston, Texas
- China (3):
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Shanghai
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061